CLINICAL TRIAL: NCT02066818
Title: Injectable Lidocaine Provides Similar Analgesia Compared to Transdermal Lidocaine/Tetracaine Patch for the Incision and Drainage of Skin Abscesses: A Randomized Controlled Trial
Brief Title: Injectable Lidocaine Versus Lidocaine/Tetracaine Patch for the Incision and Drainage of Skin Abscesses
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Christina L. Bourne, Clinical Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ECUEM-Synera
Record Dates: First submitted 2013-11-18; First posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Cutaneous Abscess; Pain
Keywords: local anesthetic; incision and drainage; pain; cutaneous abscess
MeSH Terms: conditions — Pain; Surgical Wound | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine Injection (Active Comparator): Incision and drainage performed after patient received placebo patch with injection of 1% lidocaine into the site of the abscess.
  Interventions: Drug: 1% lidocaine
- Lidocaine/tetracaine patch (Experimental): Incision and drainage performed after patient received active lidocaine/tetracaine patch and injection of 10cc of saline into site of abscess
  Interventions: Drug: Lidocaine/tetracaine patch

INTERVENTIONS:
Drug: Lidocaine/tetracaine patch
  Other Names: Synera patch
  Arms: Lidocaine/tetracaine patch
Drug: 1% lidocaine
  Arms: Lidocaine Injection

SUMMARY:
Local anesthesia used for incision and drainage of abscesses is known to be painful.

We studied the analgesia provided by a lidocaine/tetracaine patch compared to injectable lidocaine during incision and drainage (I&D) of skin abscesses.

Local injection of lidocaine provided similar analgesia compared to the lidocaine/tetracaine patch during I&D of skin abscesses in the Emergency Department. Pain at presentation and following the procedure was similar in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Skin abscess in need of incision and drainage (judged by treating physician)

Exclusion Criteria:

* Allergy to lidocaine or tetracaine
* Non-intact skin
* Unable/unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in VAS pain score over time | Immediately prior to starting I&D (Time 0); 2-5 minutes after start of I&D (Time 1); within 1 minute of completion of I&D (Time 2)
  VAS measured at each of the 3 time points noted above.

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Bourne, MD, Principal Investigator — Medical University of South Carolina